CLINICAL TRIAL: NCT03679858
Title: Platelet Antisedimentation Rate and Multiplate ex Vivo Examinations in Cerebrovascular Patients Treated With Antiplatelet Therapy and Healthy Controls
Brief Title: Platelet Antisedimentation Rate and Multiplate Exams in Patients on Antiplatelet Therapy and Controls
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Pecs (Other)
Responsible Party: Principal Investigator, Tihamér Molnár, associate professor, University of Pecs
Other Study IDs: PTE6735
Record Dates: First submitted 2018-09-18; First posted 2018-09-20 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Cerebrovascular Disorders; Platelet Refractoriness; Platelet Aggregation, Spontaneous
MeSH Terms: conditions — Cerebrovascular Disorders; Platelet Aggregation, Spontaneous | interventions — Platelet Function Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Platelet function test in patients: Platelet function test in patients on antiplatelet therapy
  Interventions: Other: Platelet function test
- Platelet function test in healthy: Platelet function test in healthy subjects
  Interventions: Other: Platelet function test

INTERVENTIONS:
Other: Platelet function test — Ex vivo platelet aggregation analysis by Multiplate aggregometer

SUMMARY:
To search for simple laboratory methods selecting patients with low/non-responsiveness to P2Y12 receptor antagonists.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent

Exclusion Criteria:

* Declined informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cerebrovascular disorders on antiplatelet therapy as a secundary prevention.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-10-01 (Estimated); Study Completion 2019-01-01 (Estimated)

PRIMARY OUTCOMES:
Major cerebrovascular event | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Tihamer Molnar, MD, PhD, Principal Investigator — University of Pécs Medical School
Locations (1):
- University of Pécs, Pécs, Baranya, Hungary

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant's aggregometry data will be shared with other researchers.

REFERENCES:
- See also: description about Multiple Electrode Aggregometry — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC5578190/pdf/ijms-18-01803.pdf